CLINICAL TRIAL: NCT01602159
Title: Revascularization With Open Bypass Versus Angioplasty and STenting of the Lower Extremity Trial (ROBUST)
Acronym: ROBUST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NA_00027939
Record Dates: First submitted 2012-05-16; First posted 2012-05-18 (Estimated); Last update posted 2018-09-28 (Actual); Status verified 2018-09

CONDITIONS: Superficial Femoral Artery Stenosis; Superficial Femoral Artery Occlusion; Claudication; Rest Pain
Keywords: Claudication; SFA; Open Bypass; Angioplasty; Stenting
MeSH Terms: conditions — Intermittent Claudication | interventions — Angioplasty; Stents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Open Bypass Surgery (Active Comparator): Open Bypass Surgery
  Interventions: Procedure: Open Bypass Surgery
- Angioplasty and Stenting (Active Comparator)
  Interventions: Procedure: Angioplasty and Stenting

INTERVENTIONS:
Procedure: Open Bypass Surgery — Open Bypass Surgery with Autogenous vein or PTFE Graft
  Arms: Open Bypass Surgery
Procedure: Angioplasty and Stenting — Angioplasty and Stenting of the superficial Femoral artery with Nitinol stent (Life Stent flexStar Stent System by Bard Inc. Tempe AZ).
  Other Names: Life Stent flexStar Stent System by Bard Inc. Tempe AZ
  Arms: Angioplasty and Stenting

SUMMARY:
This is a prospective randomized controlled trial to compare clinical improvement, cost effectiveness and patency rates between new and improved Nitinol stents and open bypass surgery in the superficial femoral artery disease.

Secondary outcomes also include comparing quality of life, re-intervention rate, mortality, morbidity and time to return to work or regular activities.

Patients with superficial femoral artery lesions will be considered. Patients with TASC II A lesions will not be randomized but treated with PTA/stenting as standard of care. Patients with TASC II B and C lesions will be prospectively randomized into either receiving open bypass or stenting.

Patients with TASC D lesions will be treated with open bypass surgery after angiography.

The investigators will collect pre-procedure, peri-procedural and clinical follow-up data on all enrolled the patients.

ELIGIBILITY:
Inclusion Criteria:

Clinical Inclusion:

1. Must be at least 18 years of age.
2. Patient has been informed of the nature of the study, and has provided written informed consent, approved by the appropriate Institutional Review Board (IRB)/Medical Ethics Committee (MEC) of the respective clinical site.
3. Symptomatic patient as evidence by IC or CLI.
4. Patient has failed maximized medical treatment and exercise program.
5. Patient has a resting ABI < 0.9 or an abnormal exercise ABI if resting ABI is normal.Patient with non-compressible arteries (ABI > 1.2) must have a TBI < 0.8.
6. Patient has a de novo or restenotic lesion(s) with > 50% stenosis documented angiographically.
7. Patient agrees to return for all required clinical contacts following study enrollment.
8. Patient has no childbearing potential or has a negative pregnancy test within one week prior to the study procedure.

Anatomical Inclusion:

1. Patient with any SFA lesion
2. At least one tibial vessel runoff with < 50% stenosis
3. Lesion starts start at least 1 cm distal to the deep femoral artery
4. Lesion end at least 3 cm above the knee joint
5. Target vessel reference diameter is > 3 mm & < 6.5 mm

Exclusion Criteria:

Clinical exclusion:

1. Known allergic reaction to anesthesia not able to overcome by medication.
2. Known allergic reaction to contrast not able to overcome by medication.
3. Known history of intolerance to study medicating including ASA, clopidogrel, or ticlopidine.
4. Bleeding disorder or refuses blood transfusion.
5. Prior stenting or bypass of SFA (prior PTA is not an exclusion criteria)
6. Unstable angina, recent MI within a month
7. Malignancy or other condition limiting life expectancy to < 5 years.
8. Renal insufficiency (serum Cr > 2.0)
9. Patient has any condition that precludes proper angiographic assessment or makes percutaneous arterial access unsafe (e.g., morbid obesity).

Anatomic Exclusion:

1. Lesion < 1 cm from origin of DFA
2. Lesion < 3 cm from the knee joint
3. Chronic total occlusion of SFA > 20cm.
4. Chronic total occlusion of CFA.
5. Proximal trifurcation occlusions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2009-07 (Actual); Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Clinical improvement | 12 Month Post Operatively
  Clinical Improvement is measured as at least 1 Rutherford category
Patency rate | 12 Month Post Operatively
  Primary, primary assisted and secondary at 6, 12 month
Cost effectiveness | 12 Month Post Operatively
  Cost Effectiveness factoring procedure and hospital admission costs

SECONDARY OUTCOMES:
Quality of Life improvement | 12 Month Post Operatively
  Improvement of quality of life measured using VQL
Re-intervention rate | 12 Month Post Operatively
Technical success of both treatment modalities | 12 Month Post Operatively
30-day operative mortality | 12 Month Post Operatively
Time to return to work and regular activities | 12 Month Post Operatively
Morbidity associated with both treatment modalities | 12 Month Post Operatively

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud B Malas, M.D., MHS, Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Johns Hopkins Bayview Medical Center, Baltimore, Maryland

REFERENCES:
- [Derived] Malas MB, Qazi U, Glebova N, Arhuidese I, Reifsnyder T, Black J, Perler BA, Freischlag JA. Design of the Revascularization With Open Bypass vs Angioplasty and Stenting of the Lower Extremity Trial (ROBUST): a randomized clinical trial. JAMA Surg. 2014 Dec;149(12):1289-95. doi: 10.1001/jamasurg.2014.369. PMID 25353642
- See also: Related Info — http://www.hopkinsmedicine.org/heart_vascular_institute/clinical_trials/vascular/robust.html